CLINICAL TRIAL: NCT07167121
Title: Etude de validité Predictive du Chelsea Critical Care Physical Assessment Tool (CPAx) Quant au Retour de l'Autonomie à la Marche 3 Mois après la Sortie de réanimation
Brief Title: Predictive Validity of the Chelsea Critical Care Physical Assessment Tool (CPAx) for Regaining Autonomy Three Months After ICU Discharge
Acronym: CPAx-Predict
Status: Recruiting | Type: Observational
Sponsor: Centre Hospitalier Intercommunal Elbeuf-Louviers-Val de Reuil (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2025-A01335-44
Record Dates: First submitted 2025-08-19; First posted 2025-09-11 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: ICU Acquired Weakness; Intensive Care Neuropathy
Keywords: ICU; Physiotherapy; ICU Acquired Weakness; CPAx; Predictive Validity; Test

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Interventional Group: Assessment of the CPAx score at ICU discharge, followed by the 6-minute walk test three months after ICU Discarge.
  Interventions: Diagnostic Test: CPAx

INTERVENTIONS:
Diagnostic Test: CPAx — Evaluation of :
  Respiratory function Cough Moving within the bed Supine to sitting on the edge of the bed Dynamic sitting Standing balance Sit to stand (starting position ≥ 90°) Transfering from bed to chair Stepping Grip strength (predicted mean for age and gender on the strongest hand)

SUMMARY:
This single-center observational study aims to explore the relationship between the CPAx score (Chelsea Critical Care Physical Assessment Tool), measured at ICU discharge, and the 6-minute walk test (6MWT) distance performed 3 months after discharge. The study targets patients who experienced prolonged mechanical ventilation and were admitted to the ICU at CHI Elbeuf-Louviers-Val-de-Reuil. Eligible participants must show signs of malnutrition, muscular weakness, or post-traumatic stress symptoms. Data collection includes the CPAx score, 6MWT distance, MRC score, and relevant clinical and demographic information. The primary objective is to determine whether the CPAx score can predict long-term functional recovery and guide post-ICU rehabilitation strategies. Participants will be evaluated during routine follow-up in the day hospital. This non-interventional study poses minimal risk to participants.

ELIGIBILITY:
Inclusion Criteria:

* Patient affiliated with, or entitled to benefit from, a French social security system.
* Patient who has received clear and comprehensive information about the study and has signed the informed consent form together with the investigator.
* Age ≥ 18 years.
* Having received at least 48 hours of invasive mechanical ventilation.
* Previous hospitalization in the intensive care unit (ICU) at CHI Elbeuf-Louviers-Val-de-Reuil.
* Prescription of physiotherapy during the ICU stay.
* Eligible for the 3-month post-ICU follow-up in the day hospital based on at least one of the following criteria:

  * Mechanical ventilation or catecholamine treatment (norepinephrine) for ≥ 5 days;
  * Weight loss ≥ 5% during hospitalization (criterion for malnutrition);
  * Significant muscle weakness (MRC score < 28/60);
  * Presence of post-traumatic stress symptoms related to ICU stay (evaluated by the psychologist).
* Ability to walk (with or without assistive devices) prior to ICU admission.

Exclusion Criteria:

* Patient not affiliated with the French national health insurance system.
* Documented pre-existing cognitive impairment likely to limit understanding of instructions and participation in functional assessments (e.g., dementia, intellectual disability, severe uncontrolled psychiatric disorder).
* History of disabling chronic neuromuscular disease (e.g., amyotrophic lateral sclerosis, myopathy, progressive chronic polyneuropathy).
* History of major pre-existing locomotor impairment preventing autonomous walking (e.g., paraplegia, uncompensated disabling arthropathy).
* Refusal to participate in the study or withdrawal of consent at any time.
* Person under legal guardianship, curatorship, or any other legal protection measure.
* Simultaneous participation in another interventional study likely to interfere with the evaluation criteria of the present study.
* Medical contraindication to performing the 6-minute walk test at 3 months (e.g., cardiovascular decompensation, acute pulmonary disease, persistent hemodynamic instability).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study targets patients who experienced prolonged mechanical ventilation and were admitted to the ICU at CHI Elbeuf-Louviers-Val-de-Reuil. Eligible participants must show signs of malnutrition, muscular weakness (icuaw), or post-traumatic stress symptoms
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Predictive validity beetween CPAx test and 6MWT | Three months after discharge
  Evaluation Criteria:
  The statistical analysis will primarily aim to assess the correlation between the CPAx score, a discrete quantitative variable (ranging from 0 to 50), and the distance covered in the 6-Minute Walk Test (6MWT), a continuous quantitative variable. The alpha risk is set at 5% and the beta risk at 80%. A sample size of 25 patients has been determined to allow for an initial estimate, accounting for an anticipated 20% loss to follow-up, in line with recommendations for feasibility studies in intensive care settings.
  Method :
  The choice of correlation test will depend on data distribution:
  * If CPAx and 6MWT distributions are normal (as verified by Shapiro-Wilk or Kolmogorov-Smirnov tests), Pearson's correlation will be used.
  * In the absence of normality or in the presence of significant skewness, Spearman's correlation (a non-parametric test) will be preferred.

SECONDARY OUTCOMES:
Correlation between CPAx and SF-36 questionnary | Three months after discharge
  Analysis of the correlation between each item of the CPAx and the results of the 6-minute walk test three months after ICU discharge.
  Analysis of the correlation between individual CPAx item scores and SF-36 questionnaire results three months after ICU discharge
  Methods for Secondary Outcomes:
  * Correlation between CPAx items and 6MWT: Each CPAx item will be analyzed individually as a discrete ordinal variable. Spearman's correlation will be used.
  * Correlation between overall CPAx score and SF-36 dimensions: These correlations will be assessed using Spearman's test, unless normality of SF-36 subscales is confirmed.
  Exploratory analyses using simple or multiple linear regression may also be conducted to model the relationship between CPAx and 6MWT, adjusting for clinical variables (age, BMI, duration of ventilation, etc.).

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Hospitalier Intercommunal Elbeuf-Louviers-Val de Reuil, Saint-Aubin-lès-Elbeuf, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Corner EJ, Soni N, Handy JM, Brett SJ. Construct validity of the Chelsea critical care physical assessment tool: an observational study of recovery from critical illness. Crit Care. 2014 Mar 27;18(2):R55. doi: 10.1186/cc13801. PMID 24669784
- [Background] Skinner EH, Thomas P, Reeve JC, Patman S. Minimum standards of clinical practice for physiotherapists working in critical care settings in Australia and New Zealand: A modified Delphi technique. Physiother Theory Pract. 2016 Aug;32(6):468-482. doi: 10.3109/09593985.2016.1145311. Epub 2016 Jun 3. PMID 27259819
- [Background] Corner EJ, Wood H, Englebretsen C, Thomas A, Grant RL, Nikoletou D, Soni N. The Chelsea critical care physical assessment tool (CPAx): validation of an innovative new tool to measure physical morbidity in the general adult critical care population; an observational proof-of-concept pilot study. Physiotherapy. 2013 Mar;99(1):33-41. doi: 10.1016/j.physio.2012.01.003. Epub 2012 Mar 30. PMID 23219649
- [Background] De Jonghe B, Bastuji-Garin S, Durand MC, Malissin I, Rodrigues P, Cerf C, Outin H, Sharshar T; Groupe de Reflexion et d'Etude des Neuromyopathies en Reanimation. Respiratory weakness is associated with limb weakness and delayed weaning in critical illness. Crit Care Med. 2007 Sep;35(9):2007-15. doi: 10.1097/01.ccm.0000281450.01881.d8. PMID 17855814
- [Background] Ali NA, O'Brien JM Jr, Hoffmann SP, Phillips G, Garland A, Finley JC, Almoosa K, Hejal R, Wolf KM, Lemeshow S, Connors AF Jr, Marsh CB; Midwest Critical Care Consortium. Acquired weakness, handgrip strength, and mortality in critically ill patients. Am J Respir Crit Care Med. 2008 Aug 1;178(3):261-8. doi: 10.1164/rccm.200712-1829OC. Epub 2008 May 29. PMID 18511703
- [Background] De Jonghe B, Sharshar T, Lefaucheur JP, Authier FJ, Durand-Zaleski I, Boussarsar M, Cerf C, Renaud E, Mesrati F, Carlet J, Raphael JC, Outin H, Bastuji-Garin S; Groupe de Reflexion et d'Etude des Neuromyopathies en Reanimation. Paresis acquired in the intensive care unit: a prospective multicenter study. JAMA. 2002 Dec 11;288(22):2859-67. doi: 10.1001/jama.288.22.2859. PMID 12472328
- [Background] Herridge MS, Cheung AM, Tansey CM, Matte-Martyn A, Diaz-Granados N, Al-Saidi F, Cooper AB, Guest CB, Mazer CD, Mehta S, Stewart TE, Barr A, Cook D, Slutsky AS; Canadian Critical Care Trials Group. One-year outcomes in survivors of the acute respiratory distress syndrome. N Engl J Med. 2003 Feb 20;348(8):683-93. doi: 10.1056/NEJMoa022450. PMID 12594312
- [Background] Latronico N, Bolton CF. Critical illness polyneuropathy and myopathy: a major cause of muscle weakness and paralysis. Lancet Neurol. 2011 Oct;10(10):931-41. doi: 10.1016/S1474-4422(11)70178-8. PMID 21939902
- [Background] Tipping CJ, Harrold M, Holland A, Romero L, Nisbet T, Hodgson CL. The effects of active mobilisation and rehabilitation in ICU on mortality and function: a systematic review. Intensive Care Med. 2017 Feb;43(2):171-183. doi: 10.1007/s00134-016-4612-0. Epub 2016 Nov 18. PMID 27864615
- See also: Rehabilitation after critical illness in adults (Clinical guideline [CG83]) — https://www.nice.org.uk/guidance/cg83
- See also: Diagnostic et prise en charge des patients adultes avec un syndrome post-réanimation (PICS) et de leur entourage — https://www.has-sante.fr/jcms/p_3445496/fr/decision-n2023-0190/dc/sbp-du-17-mai-2023